CLINICAL TRIAL: NCT00473382
Title: A Phase III, Double-masked, Multicenter, Randomized, Sham Injection-controlled Study of the Efficacy and Safety of Ranibizumab Injection in Subjects With Clinically Significant Macular Edema With Center Involvement Secondary to Diabetes Mellitus
Brief Title: A Study of Ranibizumab Injection in Subjects With Clinically Significant Macular Edema (ME) With Center Involvement Secondary to Diabetes Mellitus (RIDE)
Acronym: RIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FVF4168g
Record Dates: First submitted 2007-05-13; First posted 2007-05-15 (Estimated); Results first posted 2013-01-17 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus; Macular Edema
Keywords: Lucentis; DME; Diabetes; Vision loss
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema; Vision Disorders | interventions — Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Ranibizumab 0.3 mg (Experimental): Patients received ranibizumab 0.3 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months.
  Interventions: Drug: Ranibizumab
- Ranibizumab 0.5 mg (Experimental): Patients received ranibizumab 0.5 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months.
  Interventions: Drug: Ranibizumab
- Sham injection/ranibizumab 0.5 mg (Sham Comparator): Patients received a sham intravitreal injection monthly for 24 months. Patients who had not discontinued treatment by Month 24 could choose to receive ranibizumab 0.5 mg monthly administered intravitreally for the subsequent 12 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months.
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: Ranibizumab — Sterile solution for intravitreal injection.
  Other Names: Lucentis
  Arms: Ranibizumab 0.3 mg; Ranibizumab 0.5 mg
Drug: Sham injection
  Arms: Sham injection/ranibizumab 0.5 mg

SUMMARY:
This study is a Phase III, double-masked, multicenter, randomized, sham injection-controlled study of the efficacy and safety of ranibizumab injection in patients with clinically significant macular edema with center involvement (CSME-CI) secondary to diabetes mellitus (Type 1 or 2). This study is identical in design to study NCT00473330 (Protocol ID FVF4170g).

The open-label extension phase of the study was stopped after receiving FDA approval of the study drug (ranibizumab) for diabetic macular edema.

DETAILED DESCRIPTION:
This study is composed of 3 phases: (1) A 24-month controlled treatment period (monthly treatment with ranibizumab 0.3 mg, ranibizumab 0.5 mg, or sham injection) followed by (2) a 12-month treatment period in which patients randomized to the sham group who had not discontinued from treatment (still masked) could choose to receive monthly ranibizumab 0.5 mg while the 2 ranibizumab treatment groups continued on the same treatment they received in the first 2 years. Patients who had not discontinued treatment by Month 36 were eligible to continue treatment with ranibizumab 0.5 mg as needed (pro re nata, PRN) in (3) an extension phase of the study for up to 2 more years, resulting in up to 5 years possible total treatment time for some patients.

As per the protocol, Genentech terminated the study approximately 30 days after approval of ranibizumab for diabetic macular edema in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide written informed consent and, at U.S. sites, Health Insurance Portability and Accountability Act (HIPAA) authorization, and in other countries, as applicable according to national laws.
* Age ≥ 18 years.
* Diabetes mellitus (Type 1 or 2) .
* Retinal thickening secondary to diabetes mellitus (DME) involving the center of the fovea with central macular thickness ≥ 275 µm in the center subfield as assessed on optical coherence tomography (OCT).
* Best corrected visual acuity (BCVA) score in the study eye of 20/40 to 20/320 approximate Snellen equivalent using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at an initial testing distance of 4 meters.
* Decrease in vision determined to be primarily the result of DME and not to other causes.
* For sexually active women of childbearing potential, use of an appropriate form of contraception (or abstinence) for the duration of the study.
* Ability (in the opinion of the investigator) and willingness to return for all scheduled visits and assessments.

Exclusion Criteria:

* History of vitreoretinal surgery in the study eye.
* Panretinal photocoagulation (PRP) or macular laser photocoagulation in the study eye within 3 months of screening.
* Previous use of intraocular corticosteroids in the study eye (eg, triamcinolone acetonide [TA]) within 3 months of screening.
* Previous treatment with anti-angiogenic drugs in either eye (pegaptanib sodium, anecortave acetate, bevacizumab, ranibizumab, etc) within 3 months of the Day 0 (first day of treatment) visit.
* Proliferative diabetic retinopathy (PDR) in the study eye, with the exception of inactive, regressed PDR.
* Iris neovascularization, vitreous hemorrhage, traction retinal detachment, or preretinal fibrosis involving the macula in the study eye.

Concurrent Ocular Conditions

* Vitreomacular traction or epiretinal membrane in the study eye.
* Ocular inflammation (including trace or above) in the study eye.
* History of idiopathic or autoimmune uveitis in either eye.
* Structural damage to the center of the macula in the study eye that is likely to preclude improvement in VA following the resolution of macular edema, including atrophy of the retinal pigment epithelium (RPE), subretinal fibrosis, or organized hard-exudate plaque.
* Ocular disorders in the study eye that may confound interpretation of study results, including retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization (CNV) of any cause (eg, age-related macular degeneration (AMD), ocular histoplasmosis, or pathologic myopia).
* Concurrent disease in the study eye that would compromise visual acuity or require medical or surgical intervention during the study period.
* Cataract surgery in the study eye within 3 months, yttrium-aluminum-garnet (YAG) laser capsulotomy within the past 2 months, or any other intraocular surgery within the 90 days preceding Day 0.
* Aphakia or absence of the posterior capsule in the study eye.
* Uncontrolled glaucoma or previous filtration surgery in the study eye.
* Spherical equivalent of the refractive error in the study eye of more than -8 diopters myopia.
* Evidence at examination of infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye or current treatment for serious systemic infection.
* Uncontrolled blood pressure.
* History of cerebral vascular accident or myocardial infarction within 3 months prior to Day 0.
* Uncontrolled diabetes mellitus.
* Renal failure requiring dialysis or renal transplant.
* Participation in an investigational trial within 30 days prior to screening that involved treatment with any drug (excluding vitamins and minerals) or device.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or renders the subject at high risk from treatment complications.
* Pregnancy or lactation.
* History of allergy to fluorescein.
* History of allergy to ranibizumab injection or related molecule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2007-06; Primary Completion 2011-01 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Ehrlich, M.D., Ph.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Bressler N, Haskova Z, Kapre A, Gentile B. Clinically Meaningful Change Estimates for the National Eye Institute Visual Function Questionnaire-25 in Patients With Diabetic Macular Edema. Transl Vis Sci Technol. 2024 Dec 2;13(12):27. doi: 10.1167/tvst.13.12.27. PMID 39680390
- [Derived] Stockwell AD, Chang MC, Mahajan A, Forrest W, Anegondi N, Pendergrass RK, Selvaraj S, Reeder J, Wei E, Iglesias VA, Creps NM, Macri L, Neeranjan AN, van der Brug MP, Scales SJ, McCarthy MI, Yaspan BL. Multi-ancestry GWAS analysis identifies two novel loci associated with diabetic eye disease and highlights APOL1 as a high risk locus in patients with diabetic macular edema. PLoS Genet. 2023 Aug 16;19(8):e1010609. doi: 10.1371/journal.pgen.1010609. eCollection 2023 Aug. PMID 37585454
- [Derived] Talcott KE, Valentim CCS, Hill L, Stoilov I, Singh RP. Baseline Diabetic Retinopathy Severity and Time to Diabetic Macular Edema Resolution with Ranibizumab Treatment: A Meta-Analysis. Ophthalmol Retina. 2023 Jul;7(7):605-611. doi: 10.1016/j.oret.2023.02.003. Epub 2023 Feb 10. PMID 36774994
- [Derived] Gonzalez VH, Wang PW, Ruiz CQ. Panretinal Photocoagulation for Diabetic Retinopathy in the RIDE and RISE Trials: Not "1 and Done". Ophthalmology. 2021 Oct;128(10):1448-1457. doi: 10.1016/j.ophtha.2019.08.010. Epub 2019 Aug 21. PMID 31668888
- [Derived] Wykoff CC, Eichenbaum DA, Roth DB, Hill L, Fung AE, Haskova Z. Ranibizumab Induces Regression of Diabetic Retinopathy in Most Patients at High Risk of Progression to Proliferative Diabetic Retinopathy. Ophthalmol Retina. 2018 Oct;2(10):997-1009. doi: 10.1016/j.oret.2018.06.005. Epub 2018 Aug 1. PMID 31047503
- [Derived] Moshfeghi AA, Shapiro H, Lemmon LA, Gune S. Impact of Cataract Surgery during Treatment with Ranibizumab in Patients with Diabetic Macular Edema. Ophthalmol Retina. 2018 Feb;2(2):86-90. doi: 10.1016/j.oret.2017.05.003. Epub 2017 Jul 27. PMID 31047350
- [Derived] Sun JK, Wang PW, Taylor S, Haskova Z. Durability of Diabetic Retinopathy Improvement with As-Needed Ranibizumab: Open-Label Extension of RIDE and RISE Studies. Ophthalmology. 2019 May;126(5):712-720. doi: 10.1016/j.ophtha.2018.10.041. Epub 2018 Nov 9. PMID 30419298
- [Derived] Reddy RK, Pieramici DJ, Gune S, Ghanekar A, Lu N, Quezada-Ruiz C, Baumal CR. Efficacy of Ranibizumab in Eyes with Diabetic Macular Edema and Macular Nonperfusion in RIDE and RISE. Ophthalmology. 2018 Oct;125(10):1568-1574. doi: 10.1016/j.ophtha.2018.04.002. Epub 2018 May 8. PMID 29752001
- [Derived] Singh RP, Habbu K, Ehlers JP, Lansang MC, Hill L, Stoilov I. The Impact of Systemic Factors on Clinical Response to Ranibizumab for Diabetic Macular Edema. Ophthalmology. 2016 Jul;123(7):1581-7. doi: 10.1016/j.ophtha.2016.03.038. Epub 2016 May 24. PMID 27234930
- [Derived] Pieramici DJ, Wang PW, Ding B, Gune S. Visual and Anatomic Outcomes in Patients with Diabetic Macular Edema with Limited Initial Anatomic Response to Ranibizumab in RIDE and RISE. Ophthalmology. 2016 Jun;123(6):1345-50. doi: 10.1016/j.ophtha.2016.02.007. Epub 2016 Mar 15. PMID 26992841
- [Derived] Bressler NM, Varma R, Mitchell P, Suner IJ, Dolan C, Ward J, Ferreira A, Ehrlich JS, Turpcu A. Effect of Ranibizumab on the Decision to Drive and Vision Function Relevant to Driving in Patients With Diabetic Macular Edema: Report From RESTORE, RIDE, and RISE Trials. JAMA Ophthalmol. 2016 Feb;134(2):160-6. doi: 10.1001/jamaophthalmol.2015.4636. PMID 26584450
- [Derived] Boyer DS, Nguyen QD, Brown DM, Basu K, Ehrlich JS; RIDE and RISE Research Group. Outcomes with As-Needed Ranibizumab after Initial Monthly Therapy: Long-Term Outcomes of the Phase III RIDE and RISE Trials. Ophthalmology. 2015 Dec;122(12):2504-13.e1. doi: 10.1016/j.ophtha.2015.08.006. Epub 2015 Oct 9. PMID 26452713
- [Derived] Bansal AS, Khurana RN, Wieland MR, Wang PW, Van Everen SA, Tuomi L. Influence of Glycosylated Hemoglobin on the Efficacy of Ranibizumab for Diabetic Macular Edema: A Post Hoc Analysis of the RIDE/RISE Trials. Ophthalmology. 2015 Aug;122(8):1573-9. doi: 10.1016/j.ophtha.2015.04.029. Epub 2015 Jun 4. PMID 26050541
- [Derived] Bressler NM, Varma R, Suner IJ, Dolan CM, Ward J, Ehrlich JS, Colman S, Turpcu A; RIDE and RISE Research Groups. Vision-related function after ranibizumab treatment for diabetic macular edema: results from RIDE and RISE. Ophthalmology. 2014 Dec;121(12):2461-72. doi: 10.1016/j.ophtha.2014.07.008. Epub 2014 Aug 20. PMID 25148789
- [Derived] Campochiaro PA, Wykoff CC, Shapiro H, Rubio RG, Ehrlich JS. Neutralization of vascular endothelial growth factor slows progression of retinal nonperfusion in patients with diabetic macular edema. Ophthalmology. 2014 Sep;121(9):1783-9. doi: 10.1016/j.ophtha.2014.03.021. Epub 2014 Apr 24. PMID 24768239
- [Derived] Brown DM, Nguyen QD, Marcus DM, Boyer DS, Patel S, Feiner L, Schlottmann PG, Rundle AC, Zhang J, Rubio RG, Adamis AP, Ehrlich JS, Hopkins JJ; RIDE and RISE Research Group. Long-term outcomes of ranibizumab therapy for diabetic macular edema: the 36-month results from two phase III trials: RISE and RIDE. Ophthalmology. 2013 Oct;120(10):2013-22. doi: 10.1016/j.ophtha.2013.02.034. Epub 2013 May 22. PMID 23706949
- [Derived] Ip MS, Domalpally A, Hopkins JJ, Wong P, Ehrlich JS. Long-term effects of ranibizumab on diabetic retinopathy severity and progression. Arch Ophthalmol. 2012 Sep;130(9):1145-52. doi: 10.1001/archophthalmol.2012.1043. PMID 22965590

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from study sites in the United States, Argentina, Peru, Columbia, Chile, and Peru. There were 47 patients from the Latin American countries.
Period: Core Study
Arm/Group | Sham Injection/Ranibizumab 0.5 mg | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg
Started | 130 | 125 | 127
Completed | 102 | 98 | 98
Not Completed | 28 | 27 | 29
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Death | 3 | 5 | 10
Not completed — Lost to Follow-up | 3 | 3 | 3
Not completed — Physician Decision | 1 | 2 | 2
Not completed — Subject non-compliance | 5 | 2 | 1
Not completed — Subject needed other treatment | 1 | 3 | 2
Not completed — Subject's decision | 12 | 11 | 10
Period: Open-label Extension Through Month 48
Arm/Group | Sham Injection/Ranibizumab 0.5 mg | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg
Started | 88 (Not all participants who completed the core study entered the optional open-label extension.) | 83 (Not all participants who completed the core study entered the optional open-label extension.) | 84 (Not all participants who completed the core study entered the optional open-label extension.)
Completed | 38 | 42 | 37
Not Completed | 50 | 41 | 47
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 1 | 3 | 3
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Subject's Decision | 5 | 1 | 6
Not completed — Sponsor's Decision to Terminate Study | 41 | 34 | 36
Not completed — Subject Required Other Intervention | 2 | 1 | 0
Period: Open-label Extension Through Month 60
Arm/Group | Sham Injection/Ranibizumab 0.5 mg | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg
Started | 88 (Not all participants who completed the core study entered the optional open-label extension.) | 83 (Not all participants who completed the core study entered the optional open-label extension.) | 84 (Not all participants who completed the core study entered the optional open-label extension.)
Completed | 2 | 1 | 2
Not Completed | 86 | 82 | 82
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Death | 1 | 7 | 4
Not completed — Lost to Follow-up | 1 | 3 | 1
Not completed — Subject's Decision | 7 | 1 | 6
Not completed — Sponsor's Decision to Terminate Study | 75 | 70 | 69
Not completed — Subject Required Other Intervention | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics of the patients enrolled in the open-label extension phase (N=88, 83, 84 patients originally randomized to the ranibizumab 0.3 mg, ranibizumab 0.5 mg, and sham injection groups, respectively) were similar to the Baseline Characteristics of the patients enrolled in the core study.
Groups:
- Ranibizumab 0.3 mg: Patients randomized to this group received ranibizumab 0.3 mg monthly administered intravitreally for 24 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months.
- Ranibizumab 0.5 mg: Patients randomized to this group received ranibizumab 0.5 mg monthly administered intravitreally for 24 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months.
- Sham Injection: Patients randomized to this group received a sham intravitreal injection monthly for 24 months.
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection | Total
Number analyzed (Participants) | 125 | 127 | 130 | 382
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (11.1) | 61.8 (10.1) | 63.5 (10.8) | 62.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 47 | 64 | 163
  Male | 73 | 80 | 66 | 219

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Gained ≥ 15 Letters in Their Best Corrected Visual Acuity (BCVA) Score From Baseline at Month 24
Description: BCVA was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart starting at a test distance of 4 meters. The BCVA score is the number of letters read correctly by the patient. An increase in the BCVA score indicates an improvement of vision.
Time Frame: Baseline to Month 24
Population: Intent-to-treat population: All randomized patients, whether or not treatment was received. Missing data were imputed using the last observation carried forward.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Ranibizumab 0.3 mg: Patients randomized to this group received ranibizumab 0.3 mg monthly administered intravitreally for 24 months.
- Ranibizumab 0.5 mg: Patients randomized to this group received ranibizumab 0.5 mg monthly administered intravitreally for 24 months.
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 125 | 127 | 130
Percentage of patients | 33.6 [25.3 to 41.9] | 45.7 [37.0 to 54.3] | 12.3 [6.7 to 18.0]
Statistical Analysis 1: Comparison: Ranibizumab 0.3 mg vs Sham Injection; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — An adjustment was made for multiple treatment comparisons of the ranibizumab dose groups with the control group; The analysis was stratified by baseline BCVA score (≤55, >55 letters), baseline HbA1c (≤8%, >8%), and prior therapy for ME in the study eye (yes, no); Difference in percentage at Month 24 = 20.8, 95% CI 2-sided [11.4 to 30.2] — The percentage for each group and the difference in percentage between groups were estimated using the weighted average of the observed percentages and the differences in observed percentages over the strata using the Cochran-Mantel-Haenszel weights
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Sham Injection; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — An adjustment was made for multiple treatment comparisons of the ranibizumab dose groups with the control group; [statistical method as in outcome 1, analysis 1]; Difference in percentage at Month 24 = 33.3, 95% CI 2-sided [23.8 to 42.8] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Score at Months 24, 36, and 48
Description: BCVA was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart starting at a test distance of 4 meters. The BCVA score is the number of letters read correctly by the patient. An increase in the BCVA score indicates an improvement of vision. A positive change score indicates improvement.
Time Frame: Baseline to Month 48
Population: Intent-to-treat population: All randomized patients, whether or not treatment was received. Missing data were imputed up to Month 36 using the last observation carried forward method. The Month 48 outcome measures are based on the observed data for patients enrolled in the open-label extension phase; missing data were not imputed.
Measure: Mean (Standard Deviation); unit: Letters
Groups:
- Ranibizumab 0.3 mg: Patients randomized to this group received ranibizumab 0.3 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. For 24-month outcome measures, data in this column represents efficacy data at Month 24. For 36-month outcome measures, data in this column represents efficacy data at Month 36. For 48-month outcome measures, data in this column represents efficacy data at Month 48 for subjects enrolled in the open-label extension.
- Ranibizumab 0.5 mg: Patients randomized to this group received ranibizumab 0.5 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. For 24-month outcome measures, data in this column represents efficacy data at Month 24. For 36-month outcome measures, data in this column represents efficacy data at Month 36. For 48-month outcome measures, data in this column represents efficacy data at Month 48 for subjects enrolled in the open-label extension.
- Sham Injection: Patients randomized to this group received a sham intravitreal injection monthly for 24 months. For 24-month outcome measures, data in this column represents efficacy data at Month 24.
- Sham Injection/Ranibizumab 0.5 mg: Patients randomized to this group received a sham intravitreal injection monthly for 24 months. Although still masked, patients who had not discontinued treatment by Month 24 could choose to receive ranibizumab 0.5 mg monthly administered intravitreally for the subsequent 12 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. For 36-month outcome measures, data in this column represents efficacy data at Month 36. For 48-month outcome measures, data in this column represents efficacy data at Month 48 for subjects enrolled in the open-label extension.
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 125 | 127 | 130 | 130
Letters
  Month 24 | 10.9 (10.4) | 12.0 (14.9) | 2.3 (14.2) | NA (NA) — NA = not applicable, see reporting groups.
  Month 36 | 10.6 (12.9) | 11.4 (16.3) | NA (NA) — NA = not applicable, see reporting groups. | 4.7 (13.3)
  Month 48 (n=34,39,39,0) | 11.1 (12.0) | 12.4 (9.7) | NA (NA) — NA = not applicable, see reporting groups. | 4.6 (12.8)
Statistical Analysis 1: Comparison: Ranibizumab 0.3 mg vs Sham Injection; The analysis summarized in this section is for the Month 24 time point, comparing the outcome for patients randomized to ranibizumab versus sham injections during the controlled treatment period. The statistical analysis for the Outcome Measure at Month 36 is not shown here. The statistical analysis was not performed at Month 48; Test type: Superiority or Other; p < 0.0001, ANOVA — To manage the type I error rate while testing multiple secondary efficacy endpoints for statistical significance, a type I error management plan was implemented. Secondary endpoints were prioritized and tested using a hierarchical testing procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.5, 95% CI 2-sided [5.4 to 11.5]
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Sham Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 9.9, 95% CI 2-sided [6.4 to 13.3]

3. Secondary Outcome: Percentage of Patients With a Visual Acuity (VA) Snellen Equivalent of 20/40 or Better at Months 24, 36, and 48
Description: VA was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart starting at a test distance of 4 meters. An increase in the number of lines read correctly by the patient in the ETDRS chart indicates an improvement of vision. The Snellen equivalent of 20/40 or better is 69 or more letters correctly read in the EDTRS chart.
Time Frame: Months 24, 36, and 48
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 125 | 127 | 130 | 130
Percentage of patients
  Month 24 | 54.4 [45.7 to 63.1] | 62.2 [53.8 to 70.6] | 34.6 [26.4 to 42.8] | NA [NA to NA] — NA = not applicable, see reporting groups.
  Month 36 | 55.2 [46.5 to 63.9] | 59.1 [50.5 to 67.6] | NA [NA to NA] — NA = not applicable, see reporting groups. | 42.3 [33.8 to 50.8]
  Month 48 (n=39,39,0,34) | 64.1 [47.2 to 78.8] | 56.4 [39.6 to 72.2] | NA [NA to NA] — NA = not applicable, see reporting groups. | 47.1 [29.8 to 64.9]
Statistical Analysis 1: Comparison: Ranibizumab 0.3 mg vs Sham Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in percentage at Month 24 = 21.4, 95% CI 2-sided [10.8 to 31.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Sham Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in percentage at Month 24 = 27.1, 95% CI 2-sided [16.4 to 37.9] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Patients Who Lost < 15 Letters in Their Best Corrected Visual Acuity (BCVA) Score From Baseline at Months 24, 36, and 48
Description: as for outcome 1
Time Frame: Baseline to Month 48
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 125 | 127 | 130 | 130
Percentage of patients
  Month 24 | 98.4 [96.2 to 100.0] | 96.1 [92.7 to 99.4] | 91.5 [86.8 to 96.3] | NA [NA to NA] — NA = not applicable, see reporting groups.
  Month 36 | 96.8 [93.7 to 99.9] | 96.1 [92.7 to 99.4] | NA [NA to NA] — NA = not applicable, see reporting groups. | 92.3 [87.7 to 96.9]
  Month 48 (n=39,39,0,34) | 97.4 [86.5 to 99.9] | 97.4 [86.5 to 99.9] | NA [NA to NA] — NA = not applicable, see reporting groups. | 94.1 [80.3 to 99.3]
Statistical Analysis 1: Comparison: Ranibizumab 0.3 mg vs Sham Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0119, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in percentage at Month 24 = 7.1, 95% CI 2-sided [1.7 to 12.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Sham Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1384, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in percentage at Month 24 = 4.5, 95% CI 2-sided [-1.2 to 10.1] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Score at Months 24 and 36 in Patients With Focal Edema at Baseline
Description: as for outcome 2
Time Frame: Baseline to Month 36
Population: Subgroup of the intent-to-treat population: All randomized patients with focal edema at baseline, whether or not treatment was received. Missing data were imputed using the last observation carried forward method.
Measure: Mean (Standard Deviation); unit: Letters
Groups:
- Ranibizumab 0.3 mg: Patients randomized to this group received ranibizumab 0.3 mg monthly administered intravitreally for 36 months. For 24-month outcome measures, data in this column represents efficacy data at Month 24. For 36-month outcome measures, data in this column represents efficacy data at Month 36.
- Ranibizumab 0.5 mg: Patients randomized to this group received ranibizumab 0.5 mg monthly administered intravitreally for 36 months. For 24-month outcome measures, data in this column represents efficacy data at Month 24. For 36-month outcome measures, data in this column represents efficacy data at Month 36.
- Sham Injection/Ranibizumab 0.5 mg: Patients randomized to this group received a sham intravitreal injection monthly for 24 months. Although still masked, patients who had not discontinued treatment by Month 24 could choose to receive ranibizumab 0.5 mg monthly administered intravitreally for the subsequent 12 months. For 36-month outcome measures, data in this column represents efficacy data at Month 36.
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 44 | 37 | 42 | 42
Letters
  Month 24 | 10.5 (11.9) | 12.8 (11.0) | 1.9 (17.0) | NA (NA) — NA = not applicable, see reporting groups.
  Month 36 | 10.8 (12.1) | 10.9 (16.6) | NA (NA) — NA = not applicable, see reporting groups. | 6.6 (14.4)
Statistical Analysis 1: Comparison: Ranibizumab 0.3 mg vs Sham Injection; The analysis summarized in this section is for the Month 24 time point, comparing the outcome for patients randomized to ranibizumab versus sham injections during the controlled treatment period. The statistical analysis for the Outcome Measure at Month 36 is not shown here; Test type: Superiority or Other; p = 0.0102, ANOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.3, 95% CI 2-sided [2.0 to 14.6]
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Sham Injection; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0005, ANOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 11.2, 95% CI 2-sided [5.1 to 17.3]

6. Secondary Outcome: Mean Change From Baseline in Central Foveal Thickness at Months 24, 36, and 48
Description: Central foveal thickness was assessed in optical coherence tomographic images by the central reading center. A decrease in foveal thickness suggests a reduction in macular edema. A negative change score indicates improvement.
Time Frame: Baseline to Month 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µm
Groups:
- Ranibizumab 0.5 mg: Patients randomized to this group received ranibizumab 0.5 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive Ranibizumab 0.5 mg as needed (pro re nata. PRN) for up to 24 additional months. For 24-month outcome measures, data in this column represents efficacy data at Month 24. For 36-month outcome measures, data in this column represents efficacy data at Month 36. For 48-month outcome measures, data in this column represents efficacy data at Month 48 for subjects enrolled in the open-label extension.
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 125 | 127 | 130 | 130
µm
  Month 24 | -259.8 (169.3) | -270.7 (201.6) | -125.8 (198.3) | NA (NA) — NA = not applicable, see reporting groups.
  Month 36 | -261.8 (180.8) | -266.7 (207.8) | NA (NA) — NA = not applicable, see reporting groups. | -213.2 (193.5)
  Month 48 (n=38,39,0,33) | -251.4 (173.8) | -291.6 (200.7) | NA (NA) — NA = not applicable, see reporting groups. | -258.7 (182.3)
Statistical Analysis 1: Comparison: Ranibizumab 0.3 mg vs Sham Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -111.8, 95% CI 2-sided [-151.6 to -72.0]
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Sham Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -132.2, 95% CI 2-sided [-169.7 to -94.8]

7. Secondary Outcome: Percentage of Patients With a ≥ 3-step Worsening From Baseline in the Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale Score for Eyes at Months 24 and 36
Description: The severity of diabetic retinopathy was graded on a 10-point scale by the central reading center by comparing patient fundus photographic images with a set of standard images. 1=diabetic retinopathy (DR) severity level 10, 12 (DR absent), 2=DR severity level 14A-14C, 14Z, 15, 20 (DR questionable, microaneurysms only), 3=DR severity level 35A-35F (mild non-proliferative [NP]DR), 4=DR severity level 43A, 43B (moderate NPDR), 5=DR severity level 47A-47D (moderately severe NPDR), 6=DR severity level 53A-53E (severe NPDR), 7=DR severity level 60, 61A, 61B (mild proliferative [P]DR), 8=DR severity level 65A-65C (moderate PDR), 9=DR severity level 71A-71D (high-risk PDR), 10=DR severity level 90 (cannot grade). A lower score indicates less severe diabetic retinopathy.
Time Frame: Baseline to Month 36
Population: Intent-to-treat population: All randomized patients, whether or not treatment was received. Missing data were imputed using the last observation carried forward method.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 119 | 124 | 124
Percentage of patients
  Month 24 | 1.7 [0 to 4.1] | 0 [0 to 0] | 5.6 [1.6 to 9.7] | NA [NA to NA] — NA = not applicable, see reporting groups.
  Month 36 | 0.9 [0 to 2.5] | 0.8 [0 to 2.5] | NA [NA to NA] — NA = not applicable, see reporting groups. | 3.2 [0.1 to 6.3]
Statistical Analysis 1: Comparison: Ranibizumab 0.3 mg vs Sham Injection; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0853, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in percentage at Month 24 = -4.3, 95% CI 2-sided [-9.3 to 0.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Sham Injection; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0073, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in percentage at Month 24 = -5.8, 95% CI 2-sided [-9.8 to -1.7] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percentage of Patients With Resolution of Leakage at Month 24
Description: Resolution of leakage was defined as total area of fluorescein leakage in the central, inner, and outer subfields of the 0 Disc Area. Leakage was assessed in fluorescein angiographic images by the central reading center.
Time Frame: Baseline to Month 24
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 123 | 127 | 129
Percentage of patients | 17.1 [10.4 to 23.7] | 30.7 [22.7 to 38.7] | 2.3 [0 to 4.9]
Statistical Analysis 1: Comparison: Ranibizumab 0.3 mg vs Sham Injection; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in percentage at Month 24 = 14.0, 95% CI 2-sided [6.8 to 21.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Sham Injection; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in percentage at Month 24 = 28.3, 95% CI 2-sided [20.2 to 36.4] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Mean Number of Macular Laser Treatments From Baseline Through Months 24 and 36
Description: The need for macular laser treatment was evaluated by the masked (evaluating) physician. Macular laser was administered per protocol-specified objective and subjective criteria starting at Month 3.
Time Frame: Baseline to Month 36
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Treatments
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 125 | 127 | 130 | 130
Treatments
  Month 24 | 0.7 (1.4) | 0.3 (0.7) | 1.6 (1.6) | NA (NA) — NA = not applicable, see reporting groups.
  Month 36 | 0.9 (1.8) | 0.4 (0.9) | NA (NA) — NA = not applicable, see reporting groups. | 1.7 (1.6)
Statistical Analysis 1: Comparison: Ranibizumab 0.3 mg vs Sham Injection; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.3 to -0.5]
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Sham Injection; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-1.6 to -1.0]

10. Secondary Outcome: Percentage of Patients Who Gained ≥ 15 Letters in Their Best Corrected Visual Acuity (BCVA) Score From Baseline at Months 36 and 48
Description: as for outcome 1
Time Frame: Baseline to Month 48
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Ranibizumab 0.3 mg: Patients randomized to this group received ranibizumab 0.3 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. For 36-month outcome measures, data in this column represents efficacy data at Month 36. For 48-month outcome measures, data in this column represents efficacy data at Month 48 for subjects enrolled in the open-label extension.
- Ranibizumab 0.5 mg: Patients randomized to this group received ranibizumab 0.5 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. For 36-month outcome measures, data in this column represents efficacy data at Month 36. For 48-month outcome measures, data in this column represents efficacy data at Month 48 for subjects enrolled in the open-label extension.
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 125 | 127 | 130
Percentage of patients
  Month 36 | 36.8 [28.3 to 45.3] | 40.2 [31.6 to 48.7] | 19.2 [12.5 to 26.0]
  Month 48 (n=39,39,34) | 48.7 [32.4 to 65.2] | 41.0 [25.6 to 57.9] | 17.6 [6.8 to 34.5]

11. Secondary Outcome: Mean Change From Month 36 in Best Corrected Visual Acuity (BCVA) Score in the Study Eye at Month 48
Description: as for outcome 2
Time Frame: Month 36 to Month 48
Population: Intent-to-treat population: All randomized patients, whether or not treatment was received. The Month 48 data are based on the observed data for patients enrolled in the open-label extension phase; missing data were not imputed.
Measure: Mean (Standard Deviation); unit: Letters
Groups:
- Ranibizumab 0.3 mg: Patients randomized to this group received ranibizumab 0.3 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. For 48-month outcome measures, data in this column represents efficacy data at Month 48 for subjects enrolled in the open-label extension.
- Ranibizumab 0.5 mg: Patients randomized to this group received ranibizumab 0.5 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. For 48-month outcome measures, data in this column represents efficacy data at Month 48 for subjects enrolled in the open-label extension.
- Sham Injection/Ranibizumab 0.5 mg: Patients randomized to this group received a sham intravitreal injection monthly for 24 months. Although still masked, patients who had not discontinued treatment by Month 24 could choose to receive ranibizumab 0.5 mg monthly administered intravitreally for the subsequent 12 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. For 48-month outcome measures, data in this column represents efficacy data at Month 48 for subjects enrolled in the open-label extension.
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 39 | 39 | 34
Letters | -0.9 (8.3) | 0.3 (10.7) | -2.6 (8.8)

12. Secondary Outcome: Percentage of Patients Who Lost < 15 Letters in Their Best Corrected Visual Acuity (BCVA) Score in the Study Eye From Month 36 at Month 48
Description: as for outcome 1
Time Frame: Month 36 to Month 48
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 39 | 39 | 34
Percentage of patients | 92.3 [79.1 to 98.4] | 97.4 [86.5 to 99.9] | 88.2 [72.5 to 96.7]

13. Secondary Outcome: Mean Change From Month 36 in Central Foveal Thickness in the Study Eye at Month 48
Description: as for outcome 6
Time Frame: Month 36 to Month 48
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Ranibizumab 0.3 mg | Ranibizumab 0.5 mg | Sham Injection/Ranibizumab 0.5 mg
Number analyzed (Participants) | 38 | 39 | 33
µm | 46.1 (148.1) | 44.1 (86.3) | 9.6 (78.9)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the first day of treatment through Month 60. The sham Months 0-36 group includes patients randomized to sham. The sham Months 0-24 group includes patients who received sham during the first 24 months of the study.
Description: The adverse events tables have been updated to MedDRA version 15.1 to include safety data from the open-label extension phase. Late reported adverse events from the 36-month period have also been included.
  Safety evaluable population: All randomized patients who received at least 1 study treatment.
Groups:
- Sham Injection - Months 0-24: Patients received a sham intravitreal injection monthly for 24 months. Data in this column represent the safety data in the sham group during the first 24 months of the trial when patients were receiving only sham injections. Safety data shown here are also included in the Sham/Ranibizumab 0.5 mg - Months 0-36 column.
- Sham Injection/Ranibizumab 0.5 mg - Months 0-36: Patients received a sham intravitreal injection monthly for 24 months. Although still masked, patients who had not discontinued treatment by Month 24 could choose to receive ranibizumab 0.5 mg monthly administered intravitreally for the subsequent 12 months. Data in this column represent the safety data in the sham group during the entire 36 months of the trial; most patients crossed over to receive ranibizumab 0.5 mg monthly in the third year.
- Ranibizumab 0.3 mg - Months 0-36: Patients received ranibizumab 0.3 mg monthly administered intravitreally for 36 months.
- Ranibizumab 0.5 mg - Months 0-36: Patients received ranibizumab 0.5 mg monthly administered intravitreally for 36 months.
- Sham Injection/Ranibizumab 0.5 mg - Months 37-60: Patients received a sham intravitreal injection monthly for 24 months. Although still masked, patients who had not discontinued treatment by Month 24 could choose to receive ranibizumab 0.5 mg monthly administered intravitreally for the subsequent 12 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. Data in this column represent the safety data during the open-label extension phase (after Month 36).
- Ranibizumab 0.3 mg - Months 37-60: Patients received ranibizumab 0.3 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. Data in this column represent the safety data during the open-label extension phase (after Month 36).
- Ranibizumab 0.5 mg - Months 37-60: Patients received ranibizumab 0.5 mg monthly administered intravitreally for 36 months. Patients who had not discontinued treatment by Month 36 could enter the open-label extension phase to receive ranibizumab 0.5 mg as needed (pro re nata [PRN]) for up to 24 additional months. Data in this column represent the safety data during the open-label extension phase (after Month 36).
Arm/Group | Sham Injection - Months 0-24 | Sham Injection/Ranibizumab 0.5 mg - Months 0-36 | Ranibizumab 0.3 mg - Months 0-36 | Ranibizumab 0.5 mg - Months 0-36 | Sham Injection/Ranibizumab 0.5 mg - Months 37-60 | Ranibizumab 0.3 mg - Months 37-60 | Ranibizumab 0.5 mg - Months 37-60
Serious Adverse Events (participants affected / at risk) | 54/127 | 68/127 | 54/125 | 67/124 | 19/88 | 31/83 | 18/84
Other Adverse Events (participants affected / at risk) | 123/127 | 123/127 | 120/125 | 121/124 | 65/88 | 63/83 | 62/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection - Months 0-24 (N=127) | Sham Injection/Ranibizumab 0.5 mg - Months 0-36 (N=127) | Ranibizumab 0.3 mg - Months 0-36 (N=125) | Ranibizumab 0.5 mg - Months 0-36 (N=124) | Sham Injection/Ranibizumab 0.5 mg - Months 37-60 (N=88) | Ranibizumab 0.3 mg - Months 37-60 (N=83) | Ranibizumab 0.5 mg - Months 37-60 (N=84)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 4 | 1 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 3 | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 3 | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 3 | 0 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 6 | 7 | 3 | 4 | 5 | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 3 | 2 | 6 | 0 | 2 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basedow's disease (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angle closure glaucoma (S) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — (S)=study eye
Blindness unilateral (F) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — (F)=fellow eye
Cataract (S) (Eye disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 — (S)=study eye
Choroidal neovascularisation (S) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — (S)=study eye
Corneal opacity (S) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — (S)=study eye
Diabetic retinal oedema (S) (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — (S)=study eye
Glaucoma (F) (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 — (F)=fellow eye
Macular ischaemia (F) (Eye disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 — (F)=fellow eye
Macular oedema (F) (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 — (F)=fellow eye
Macular oedema (S) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — (S)=study eye
Papilloedema (F) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — (F)=fellow eye
Retinal detachment (F) (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 — (F)=fellow eye
Retinal haemorrhage (S) (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 — (S)=study eye
Visual acuity reduced (F) (Eye disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 0 — (F)=fellow eye
Visual acuity reduced (S) (Eye disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 0 — (S)=study eye
Vitreous haemorrhage (F) (Eye disorders) | 2 | 3 | 10 | 4 | 0 | 0 | 0 — (F)=fellow eye
Appendiceal mucocoele (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 3 | 3 | 2 | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Empyema (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Endophthalmitis (F) (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — (F)=fellow eye
Endophthalmitis (S) (Infections and infestations) | 0 | 0 | 3 | 2 | 0 | 0 | 0 — (S)=study eye
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 5 | 1 | 8 | 2 | 1 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Sepsis syndrome (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract traumatic (S) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 — (S)=study eye
Corneal abrasion (S) (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 — (S)=study eye
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Expired drug administered (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 2 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0 | 0 | 1
Medication error (S) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — (S)=study eye
Post procedural complication (S) (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — (S)=study eye
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural complication (S) (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — (S)=study eye
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Intraocular pressure increased (S) (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — (S)=study eye
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 1 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 3 | 4 | 0 | 2 | 2
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 3 | 1 | 1 | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 4 | 3 | 4 | 1 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 2 | 2 | 1 | 1 | 3 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 2 | 2 | 3 | 0 | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephroureterectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 3 | 1 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vascular insufficiency (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (S) (Eye disorders) | 3 | 4 | 1 | 0 | 0 | 1 | 1 — (S)=study eye
Retinal detachment (S) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 — (S)=study eye
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 6 | 7 | 8 | 3 | 0 | 3 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endocarditis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stent placement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal vein occlusion (F) (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection - Months 0-24 (N=127) | Sham Injection/Ranibizumab 0.5 mg - Months 0-36 (N=127) | Ranibizumab 0.3 mg - Months 0-36 (N=125) | Ranibizumab 0.5 mg - Months 0-36 (N=124) | Sham Injection/Ranibizumab 0.5 mg - Months 37-60 (N=88) | Ranibizumab 0.3 mg - Months 37-60 (N=83) | Ranibizumab 0.5 mg - Months 37-60 (N=84)
Anaemia (Blood and lymphatic system disorders) | 13 | 16 | 13 | 22 | 3 | 2 | 3
Atrial fibrillation (Cardiac disorders) | 4 | 7 | 4 | 4 | 2 | 3 | 1
Cardiac failure congestive (Cardiac disorders) | 7 | 8 | 7 | 3 | 0 | 2 | 2
Coronary artery disease (Cardiac disorders) | 4 | 8 | 6 | 4 | 2 | 0 | 1
Cataract (F) (Eye disorders) | 29 | 32 | 38 | 41 | 5 | 1 | 3 — (F)=fellow eye
Cataract (S) (Eye disorders) | 35 | 39 | 31 | 35 | 5 | 6 | 5 — (S)=study eye
Cataract cortical (F) (Eye disorders) | 5 | 8 | 10 | 3 | 0 | 1 | 0 — (F)=fellow eye
Cataract cortical (S) (Eye disorders) | 5 | 6 | 8 | 5 | 3 | 2 | 1 — (S)=study eye
Cataract nuclear (F) (Eye disorders) | 1 | 2 | 10 | 5 | 0 | 1 | 0 — (F)=fellow eye
Cataract nuclear (S) (Eye disorders) | 3 | 4 | 6 | 8 | 1 | 1 | 1 — (S)=study eye
Cataract subcapsular (F) (Eye disorders) | 3 | 3 | 7 | 8 | 0 | 1 | 0 — (F)=fellow eye
Conjunctival haemorrhage (F) (Eye disorders) | 3 | 11 | 8 | 14 | 3 | 2 | 5 — (F)=fellow eye
Conjunctival haemorrhage (S) (Eye disorders) | 40 | 45 | 54 | 63 | 7 | 4 | 6 — (S)=study eye
Diabetic retinal oedema (F) (Eye disorders) | 19 | 20 | 25 | 16 | 2 | 0 | 1 — (F)=fellow eye
Diabetic retinal oedema (S) (Eye disorders) | 8 | 8 | 8 | 3 | 1 | 1 | 3 — (S)=study eye
Diabetic retinopathy (F) (Eye disorders) | 5 | 5 | 8 | 10 | 0 | 2 | 0 — (F)=fellow eye
Dry eye (F) (Eye disorders) | 8 | 10 | 5 | 8 | 5 | 2 | 1 — (F)=fellow eye
Dry eye (S) (Eye disorders) | 6 | 8 | 8 | 9 | 4 | 3 | 1 — (S)=study eye
Eye irritation (S) (Eye disorders) | 4 | 6 | 8 | 7 | 1 | 1 | 2 — (S)=study eye
Eye pain (S) (Eye disorders) | 10 | 12 | 14 | 18 | 0 | 3 | 1 — (S)=study eye
Foreign body sensation in eyes (S) (Eye disorders) | 7 | 8 | 10 | 4 | 1 | 1 | 1 — (S)=study eye
Lacrimation increased (S) (Eye disorders) | 4 | 6 | 7 | 5 | 0 | 1 | 0 — (S)=study eye
Macular fibrosis (F) (Eye disorders) | 5 | 6 | 13 | 9 | 1 | 1 | 1 — (F)=fellow eye
Macular fibrosis (S) (Eye disorders) | 11 | 14 | 7 | 8 | 4 | 1 | 3 — (S)=study eye
Macular oedema (F) (Eye disorders) | 28 | 37 | 46 | 53 | 10 | 8 | 9 — (F)=fellow eye
Macular oedema (S) (Eye disorders) | 26 | 33 | 32 | 26 | 9 | 6 | 9 — (S)=study eye
Ocular hyperaemia (S) (Eye disorders) | 10 | 10 | 5 | 5 | 0 | 1 | 1 — (S)=study eye
Posterior capsule opacification (S) (Eye disorders) | 4 | 6 | 7 | 5 | 0 | 1 | 1 — (S)=study eye
Retinal exudates (F) (Eye disorders) | 16 | 18 | 23 | 21 | 0 | 2 | 1 — (F)=fellow eye
Retinal exudates (S) (Eye disorders) | 15 | 19 | 22 | 20 | 2 | 3 | 4 — (S)=study eye
Retinal haemorrhage (F) (Eye disorders) | 20 | 31 | 32 | 40 | 6 | 9 | 8 — (F)=fellow eye
Retinal haemorrhage (S) (Eye disorders) | 22 | 26 | 22 | 34 | 4 | 9 | 7 — (S)=study eye
Retinal neovascularisation (F) (Eye disorders) | 10 | 13 | 13 | 14 | 3 | 1 | 3 — (F)=fellow eye
Retinal neovascularisation (S) (Eye disorders) | 7 | 8 | 1 | 1 | 0 | 1 | 1 — (S)=study eye
Vision blurred (S) (Eye disorders) | 5 | 5 | 10 | 5 | 1 | 2 | 0 — (S)=study eye
Vitreous detachment (F) (Eye disorders) | 19 | 20 | 13 | 12 | 1 | 3 | 1 — (F)=fellow eye
Vitreous detachment (S) (Eye disorders) | 19 | 22 | 14 | 23 | 2 | 2 | 1 — (S)=study eye
Vitreous floaters (F) (Eye disorders) | 7 | 8 | 3 | 6 | 2 | 3 | 4 — (F)=fellow eye
Vitreous floaters (S) (Eye disorders) | 4 | 6 | 10 | 13 | 4 | 1 | 3 — (S)=study eye
Vitreous haemorrhage (F) (Eye disorders) | 12 | 16 | 18 | 14 | 5 | 4 | 3 — (F)=fellow eye
Vitreous haemorrhage (S) (Eye disorders) | 16 | 17 | 3 | 4 | 2 | 3 | 1 — (S)=study eye
Constipation (Gastrointestinal disorders) | 7 | 9 | 14 | 9 | 2 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 3 | 11 | 1 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 6 | 6 | 10 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 14 | 16 | 14 | 10 | 3 | 4 | 2
Vomiting (Gastrointestinal disorders) | 9 | 10 | 6 | 7 | 0 | 1 | 2
Oedema peripheral (General disorders) | 4 | 4 | 9 | 8 | 4 | 2 | 0
Drug hypersensitivity (Immune system disorders) | 6 | 7 | 2 | 1 | 0 | 0 | 2
Seasonal allergy (Immune system disorders) | 5 | 6 | 12 | 9 | 1 | 2 | 0
Bronchitis (Infections and infestations) | 4 | 6 | 8 | 12 | 0 | 2 | 1
Cellulitis (Infections and infestations) | 4 | 9 | 5 | 4 | 2 | 0 | 0
Influenza (Infections and infestations) | 7 | 9 | 10 | 13 | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 6 | 10 | 16 | 13 | 4 | 3 | 3
Pneumonia (Infections and infestations) | 4 | 6 | 5 | 8 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 12 | 14 | 9 | 14 | 4 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 12 | 14 | 12 | 13 | 3 | 3 | 2
Urinary tract infection (Infections and infestations) | 19 | 24 | 13 | 17 | 2 | 5 | 3
Corneal abrasion (S) (Injury, poisoning and procedural complications) | 6 | 8 | 7 | 4 | 1 | 0 | 0 — (S)=study eye
Fall (Injury, poisoning and procedural complications) | 3 | 8 | 10 | 2 | 1 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 7 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 5 | 6 | 8 | 5 | 1 | 1 | 0
Blood glucose increased (Investigations) | 8 | 9 | 10 | 9 | 1 | 1 | 1
Intraocular pressure increased (F) (Investigations) | 6 | 7 | 7 | 12 | 2 | 1 | 1 — (F)=fellow eye
Intraocular pressure increased (S) (Investigations) | 14 | 17 | 20 | 25 | 2 | 2 | 3 — (S)=study eye
Diabetes mellitus (Metabolism and nutrition disorders) | 22 | 25 | 19 | 22 | 5 | 6 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 8 | 13 | 4 | 2 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 4 | 5 | 8 | 2 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 4 | 7 | 6 | 2 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 7 | 5 | 2 | 3 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 14 | 5 | 9 | 0 | 0 | 2
Diabetic neuropathy (Nervous system disorders) | 4 | 6 | 7 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 5 | 5 | 7 | 1 | 3 | 1
Headache (Nervous system disorders) | 7 | 10 | 10 | 7 | 0 | 4 | 0
Neuropathy peripheral (Nervous system disorders) | 4 | 6 | 9 | 4 | 2 | 2 | 1
Anxiety (Psychiatric disorders) | 8 | 8 | 6 | 3 | 1 | 2 | 2
Renal failure (Renal and urinary disorders) | 7 | 7 | 5 | 12 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 17 | 10 | 2 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 3 | 1 | 2 | 1 | 1
Hypertension (Vascular disorders) | 31 | 35 | 33 | 38 | 5 | 3 | 3
Hypothyroidism (Endocrine disorders) | 5 | 7 | 2 | 4 | 1 | 0 | 0
Blood urea increased (Investigations) | 5 | 6 | 8 | 5 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.